CLINICAL TRIAL: NCT05761808
Title: In Patients With Chronic Low Back Pain, Ultrasonographic Evaluation Of The Effect Of Applied Neuromuscular Electrical Stimulation In Addition To Lumber Stabilization Exercises On The Multifidus Muscle Thickness
Brief Title: Effect Of Applied Neuromuscular Electrical Stimulation In Addition To Lumber Stabilization Exercises On The Multifidus Muscle Thickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2259
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Low Back Pain
Keywords: multifidus; ultrasound
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): Lumbar stabilization exercises constitute the first step of treatment in chronic low back pain.
  Interventions: Other: exercises
- NMES Group (Active Comparator): NMES will be applied in addition to lumbar stabilization exercises.
  Interventions: Other: neuromuscular electrical stimulation

INTERVENTIONS:
Other: exercises — Before being included in the study, the multifudus muscle thickness at the L4-L5 level of each patient will be measured ultrasonographically. First of all, exercises to learn transversus abdominis activation will be performed in patients. They will then be included in the stretching and strengthening exercise program. Stretching and strengthening exercises were planned as dynamic abdominal bracing, finding and maintaining neutral position, and exercises on all fours. Exercise therapy will be applied by the same physiotherapist 3 days a week for 5 weeks. Patients will continue to exercise for 7 more weeks as a home program. During this period, they will be called once a week by phone.
  Arms: Exercise Group
Other: neuromuscular electrical stimulation — NMES intensity will be planned individually according to the patients. Before being included in the study, the multifudus muscle thickness at the L4-L5 level of each patient will be measured ultrasonographically. NMES application will be applied by a specialist physiotherapist 3 days a week for 5 weeks, for a total of 15 sessions. Exercises will be applied 3 days a week for 5 weeks, accompanied by a physiotherapist. Patients will continue to exercise for 7 more weeks as a home program. In this process, patients will be called once a week by phone.
  Arms: NMES Group

SUMMARY:
The goal of this clinical trial is to show the additive effects of neuromuscular electrical stimulation (NMES) applied to the multifidus muscle in addition to stabilization exercises in patients with chronic low back pain. The main question it aims to answer is:

* Does NMES have additional effects on multifidus muscle thickness? Participants will go under a treatment protocol combination of lumber stabilization exercises and NMES.

Researchers will compare the groups Group 1 which has only lumber stabilization exercises and Group 2 which has both exercises and NMES to see if any changes occur in multifidus muscle thickness.

DETAILED DESCRIPTION:
Chronic low back pain is defined as low back pain lasting more than 3 months. Even if the acute pathology causing the pain is treated, chronic low back pain lasting up to 1 year can be seen in 20% of the patients. 80% of the population suffers from chronic low back pain at least once in their life. The causes of chronic low back pain can be very variable. Studies show that 70% of these pains are idiopathic and non-specific, that is, due to lumbar sprain and strain. This is followed by mechanical causes with 27%; spondylosis, spinal stenosis, lumbar disc herniation, osteoporotic fractures, congenital diseases. Apart from these, 2% referred pain; Pain due to malignancy and infection is seen in 1%.

Although the aim of the treatment of chronic low back pain varies according to the patient, the main purpose is to reduce the patient's pain and improve their functions. For this purpose, many treatment programs can be given to the patient. Exercises, physical therapy modalities, pharmacological treatments and surgical methods can be used.

Lumbar stabilization exercises are exercises for the abdominal and dorsal muscles, and many studies have previously shown their positive effects on pain and disability. However, these effects are usually short-term. Therefore, combining stabilization exercises with neuromuscular electrical stimulation (NMES) in patients with chronic low back pain and its clinical effect was questioned. Although this study could not prove the additive effect of NMES statistically, it showed important results on NMES tolerance of patients with chronic low back pain.

Multifudus muscle thickness was measured ultrasonographically in the studies. These studies show that multifidus muscle thickness is reduced in patients with chronic low back pain. Multifidus thickness measurement can be done statically and dynamically with the help of ultrasonography. In a study, static and dynamic multifudus thickness measurements were made at 3 levels (L3-L4, L4-L5, L5-S1), and high reliable results were obtained at L3-L4 and L4-L5 levels, and average reliable results were obtained at L5-S1 levels in static measurements. In dynamic measurements, reliable results were not obtained at all 3 levels.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain persist more than 3 months
* NRS scale is above 3
* Agree to participation and fill in the consent form

Exclusion Criteria:

* radiculopathy
* low back pain persists less than 3 months
* neurological disease
* history of lumber spinal surgery
* pregnancy
* active skin infection
* obesity and morbid obesity (BMI more than 30)
* NMES contraindication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
multifudus muscle thickness | 3 months
  A curve probe is used for ultrasound imaging. Patients are placed prone on the examination table. A pillow is placed under the abdomen to keep the lumbosacral junction angle below 10 degrees. After visualizing the L4 spinous process in the parasagittal plane, the L4-L5 facet joint is seen by moving 2 cm laterally from the midline. Probe angulation is done to get a clearer image.

SECONDARY OUTCOMES:
low back pain change | 3 months
  Numeric rating scale (NRS) is used to convert some values that cannot be measured numerically to numeric. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end, and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.

OTHER OUTCOMES:
Oswestry disability index | 3 months
  It was developed to evaluate the degree of loss of function in low back pain. The Turkish validity and reliability of the Oswestry Disability Index (OSI), which was demonstrated in 2004, consists of 10 items. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, the degree of change in pain, travel and social life. Under each item, there are six statements that the patient marked as appropriate for his/her condition. The first statement is scored as "0" and the sixth statement is scored as "5". When the total score is calculated, it is multiplied by two and expressed as a percentage. The maximum score is "100", the minimum score is "0". As the total score increases, the level of disability also increases.
EQ- 5D- 3L General Quality of Life Scale | 3 months
  It was developed to assess health-related quality of life. It consists of two parts. The first part defines the health profile in 5 dimensions: mobility, self-care, social life, pain and psychological state. Contains 3 phrases, all according to difficulty. It is evaluated as 1: little, 2: medium, 3: too much of a problem. The second part includes the analogue scale in which individuals evaluate their current health status between 0-100.
Hospital Anxiety and Depression Scale (HAD) | 3 months
  It is a self-assessment scale developed to determine the risk of anxiety and depression in patients with physical illness and those applying to primary health care services, and to measure the level and change in severity.
Fear Avoidance Beliefs Questionnaire | 3 months
  This questionnaire is a questionnaire that measures fear avoidance beliefs evaluating the effects of physical activity and work on low back pain. The questionnaire is filled by the patient. It consists of two parts. The first part is Physical Activity consisting of 5 items, and the second part is a questionnaire collected under the title of Job consisting of 11 items. Physical Activity section can get a minimum of 0 and a maximum of 24 points. The division of labor can get a minimum of 0 and a maximum of 42 points. It is accepted that there is a decrease in fear-avoidance behavior within the department as the total score approaches 0 in the evaluation, and an increase in fear-avoidance behavior as it approaches the maximum score.
International Physical Activity Questionnaire (IPAQ) | 3 months
  The IPAQ scale was developed in order to make physical activity inadequacy a general health problem, to require large population studies and to make comparisons between countries. In a multi-country validity and reliability study, this questionnaire was shown to be at least as good as other established measures of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: emre ata, Ass. Prof., Study Director — Sultan 2. Abdulhamid Han Training and Research Hospital
Locations (1):
- Sultan 2. Abdulhamıd Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No